CLINICAL TRIAL: NCT04989374
Title: Regulation of Vitamin D Metabolism by Washed Microbiota Transplantation in Patients With Inflammatory Bowel Disease
Brief Title: Regulation of Vitamin D Metabolism by Washed Microbiota Transplantation in Patients With IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: WMT-CN-160301
Record Dates: First submitted 2021-07-22; First posted 2021-08-04 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-06

CONDITIONS: IBD
Keywords: IBD; vitaminD; WMT; microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CD patients treated with WMT: the gastrointestinal experts decided the treatment plan according to the patient's condition and the patient's wishes, these CD patients treated with WMT
- CD patients treated without WMT: the gastrointestinal experts decided the treatment plan according to the patient's condition and the patient's wishes, these CD patients treated without WMT
- UC patients treated with WMT: the gastrointestinal experts decided the treatment plan according to the patient's condition and the patient's wishes, these UC patients treated with WMT
- UC patients treated without WMT: the gastrointestinal experts decided the treatment plan according to the patient's condition and the patient's wishes, these UC patients treated without WMT

SUMMARY:
WMT could effectively induce clinical response and maintain remission in patients with Inflammatory bowel disease (IBD). VD maintains gut microbiota and gut microbiota alter intestinal vitamin D metabolism (VDM),The aim of this study was to evaluate the effect of WMT on VD metabolism by measuring the level of serum 25(OH)D in IBD patients before and after treatment

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic, relapsing disorder that is represented by Crohn's disease (CD) and Ulcerative colitis (UC), the pathogenesis of IBD is not completely understood, but it is now acknowledged that it is related to intestinal microbiota. The gut microbiota is a central regulator of host metabolism, More and more evidences show that the gut microbiota plays an important physiological role in the pathogenesis of a variety of human metabolic, immune and neurological diseases, including IBD. Fecal microbiota transplantation (FMT) transplants the gut microbiota of healthy donors into the patients' intestines, This is an effective strategy to restore the intestinal microbiota and it is also a hot research topic in recent years. Our previous studies and other studies have proved that FMT could effectively induce clinical response and maintain remission in patients with IBD. Washed microbiota transplantation (WMT) is a fecal bacteria transplantation based on Intelligent fecal bacteria separation system and strict quality control of washing process, It is a new stage of FMT development, our group have proved that WMT is safer, more precise and more quality-controllable than the crude FMT by manual.

Vitamin D(VD) has been shown to have multifaced effects on the skeletal environment,immune system and infection. A number of diseases, including tumors, Type I diabetes, IBD and autoimmune diseases are associated with VD deficiency, VD could have an important role in the prevention and possible treatment of these conditions. Several studies have shown that intestinal microbiota is closely related to VD，VD maintains gut microbiota and gut microbiota alter intestinal vitamin D metabolism (VDM). A clinical trial shows that probiotics supplementation can change the level of 25 hydroxyvitaminD(25(OH)D). Serum 25(OH)D correlates with overall storage of VD, which is the preferred clinical measure to assess VD sufficiency. The aim of this study was to evaluate the effect of WMT on VD metabolism by measuring the level of serum 25(OH)D in IBD patients before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* IBD patients aged 16-65years

Exclusion Criteria:

* previous history of partial small bowel resection;
* Abnormal thyroid and parathyroid function;
* Complicated with complicated intestinal fistula and severe infection and treated with antibiotics
* Women during pregnancy, lactation and oral contraceptives.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with UC or CD were recruited from the Second Affiliated Hospital of Nanjing Medical University between March 2016 and June 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes of vitamin D levels in IBD patients after FMT treatment | 3 months
  After WMT treatment, the level of vitamin d in IBD patients increased

CONTACTS AND LOCATIONS:
Locations (1):
- The Secon affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pickard JM, Zeng MY, Caruso R, Nunez G. Gut microbiota: Role in pathogen colonization, immune responses, and inflammatory disease. Immunol Rev. 2017 Sep;279(1):70-89. doi: 10.1111/imr.12567. PMID 28856738
- [Background] Pittayanon R, Lau JT, Yuan Y, Leontiadis GI, Tse F, Surette M, Moayyedi P. Gut Microbiota in Patients With Irritable Bowel Syndrome-A Systematic Review. Gastroenterology. 2019 Jul;157(1):97-108. doi: 10.1053/j.gastro.2019.03.049. Epub 2019 Mar 30. PMID 30940523
- [Background] Ni J, Wu GD, Albenberg L, Tomov VT. Gut microbiota and IBD: causation or correlation? Nat Rev Gastroenterol Hepatol. 2017 Oct;14(10):573-584. doi: 10.1038/nrgastro.2017.88. Epub 2017 Jul 19. PMID 28743984
- [Background] Kim JH, Kim K, Kim W. Gut microbiota restoration through fecal microbiota transplantation: a new atopic dermatitis therapy. Exp Mol Med. 2021 May;53(5):907-916. doi: 10.1038/s12276-021-00627-6. Epub 2021 May 20. PMID 34017060
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Background] Lopez-Munoz P, Beltran B, Saez-Gonzalez E, Alba A, Nos P, Iborra M. Influence of Vitamin D Deficiency on Inflammatory Markers and Clinical Disease Activity in IBD Patients. Nutrients. 2019 May 11;11(5):1059. doi: 10.3390/nu11051059. PMID 31083541
- [Background] Fletcher J, Cooper SC, Ghosh S, Hewison M. The Role of Vitamin D in Inflammatory Bowel Disease: Mechanism to Management. Nutrients. 2019 May 7;11(5):1019. doi: 10.3390/nu11051019. PMID 31067701
- [Background] Thomas RL, Jiang L, Adams JS, Xu ZZ, Shen J, Janssen S, Ackermann G, Vanderschueren D, Pauwels S, Knight R, Orwoll ES, Kado DM. Vitamin D metabolites and the gut microbiome in older men. Nat Commun. 2020 Nov 26;11(1):5997. doi: 10.1038/s41467-020-19793-8. PMID 33244003
- [Background] Jones ML, Martoni CJ, Prakash S. Oral supplementation with probiotic L. reuteri NCIMB 30242 increases mean circulating 25-hydroxyvitamin D: a post hoc analysis of a randomized controlled trial. J Clin Endocrinol Metab. 2013 Jul;98(7):2944-51. doi: 10.1210/jc.2012-4262. Epub 2013 Apr 22. PMID 23609838